CLINICAL TRIAL: NCT06237439
Title: Sharing HaRT in New Expanses: Evaluating the Move With HaRT Intervention on Improving Mental Health of Human Trafficking Survivors
Brief Title: Sharing HaRT in New Expanses
Acronym: SHiNE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: Innovations for Poverty Action (Other)
Responsible Party: Principal Investigator, Catherine Carlson, Associate Professor, University of Alabama, Tuscaloosa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-02-6355
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Depressive Symptoms; Trauma, Psychological; Anxiety Generalized
MeSH Terms: conditions — Depression; Psychological Trauma; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will not be informed of the arm of participants prior to conducting assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Move with HaRT (Experimental): Move with HaRT is a 12-session, weekly, manualized mental health intervention led by trained paraprofessionals. It is delivered in groups of 8-12 individuals and includes breathwork, yoga poses, guided meditations, and discussions aligned with weekly themes. Group discussions include topics such as noticing how we feel in our bodies, recognizing and allowing all emotions, practicing self-acceptance, and developing deeper connections with others with whom we feel safe.
  Interventions: Behavioral: Move with HaRT
- Services as Usual (Active Comparator): Services as usual are ongoing activities provided by anti-trafficking agencies that include basic counseling, vocational training, games and entertainment (e.g., movies and social activities).
  Interventions: Behavioral: Move with HaRT

INTERVENTIONS:
Behavioral: Move with HaRT — Move with HaRT is a group-based, manualized mind-body intervention.

SUMMARY:
The goal of this parallel cluster randomized control (CRT) trial is to evaluate a group-based mind-body intervention (Move with HaRT) in survivors of human trafficking. The main study aims are:

1. Determine effectiveness of the Move with HaRT intervention on PTSD, depression, and anxiety symptoms among survivors of human trafficking in Uganda
2. Explore participant characteristics (e.g., age, trafficking history, food security) that may moderate the intervention effectiveness.
3. Understand potential barriers and facilitators to future implementation and scale-up.

Participants will complete:

* Complete three surveys (baseline, endline, and 3 month follow-up)
* Participate in either Services as Usual or Move with HaRT groups
* Qualitative in-depth interviews

Researchers will compare Move with HaRT with Services as Usual to see effects on mental health symptoms.

DETAILED DESCRIPTION:
Despite significant mental health challenges experienced by human trafficking survivors, a lack of research on effective interventions exists. The proposed parallel cluster randomized control trial aims to evaluate the mental health impact of Move with HaRT with human trafficking survivors in Uganda. Move with HaRT is a group-based intervention facilitated by paraprofessionals that includes breathwork, yoga poses, meditation, and discussions. The proposed study will use a parallel cluster randomized control (CRT) trial with 302 survivors randomized in groups to either Move with HaRT or Services as Usual. The main study aims are: 1) Determine effectiveness of the Move with HaRT intervention on PTSD, depression, and anxiety symptoms among survivors of human trafficking in Uganda; 2) Explore participant characteristics (e.g., age, trafficking history, food security) that may moderate the intervention effectiveness; 3) Understand potential barriers and facilitators to future implementation and scale-up. Surveys at baseline, endline, and 3-month follow-up assess mental health outcomes, as well as secondary outcomes on physical and social wellbeing. Qualitative research will inform barriers and facilitators to future implementation and scale-up. Results of this study have the potential to inform protection services in Uganda and beyond.

ELIGIBILITY:
Inclusion Criteria:

* identify as female;
* history of forced labor or sex trafficking;
* aged 14 and above;

Exclusion Criteria:

* physically unable to perform basic day-to-day activities without assistance
* does not provide consent (or assent if a minor)

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Past two weeks
  Severity of depressive symptoms
PTSD Checklist (PCL-5) | Past one month
  Severity of post-traumatic stress symptoms
GAD-7 | Past one month
  Severity of generalized anxiety symptoms

SECONDARY OUTCOMES:
Brief Pain Inventory (Short Form) | 24 hours
  Severity of pain
Women's Health Initiative Insomnia Rating Scale (WHIIRS) | Past four weeks
  Severity of insomnia symptoms
Multidimensional Scale of Perceived Social Support (MSPSS) | Past three months
  Degree of perceived social support

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Carlson, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Innovations for Poverty Action, Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No